CLINICAL TRIAL: NCT03734471
Title: Use of a Novel Chest Tube Insertion Device for Urgent Thoracostomy in an Emergency Department Setting
Brief Title: Reactor Thoracostomy
Acronym: UNCUT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Crozer-Keystone Health System (Other)
Responsible Party: Principal Investigator, Richard Pescatore, Director of Clinical Research, Crozer-Keystone Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-025; NCT03769727 (obsolete NCT alias)
Record Dates: First submitted 2018-11-06; First posted 2018-11-08 (Actual); Last update posted 2018-11-08 (Actual); Status verified 2018-11

CONDITIONS: Pneumothorax; Hemothorax
MeSH Terms: conditions — Pneumothorax; Hemothorax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Traditional (Active Comparator)
  Interventions: Procedure: Tube thoracostomy
- Reactor Device (Experimental)
  Interventions: Device: Reactor Device

INTERVENTIONS:
Device: Reactor Device — The Reactor is a Class II FDA medical device to facilitate the insertion of chest tubes into the thoracic cavity.
  Arms: Reactor Device
Procedure: Tube thoracostomy — Traditional chest tube placement
  Arms: Traditional

SUMMARY:
Tube thoracostomy is commonly performed in the emergency department for patients suffering from traumatic hemo- or pneumo-thorax. The procedure involves the use of a scalpel incision at the skin followed by blunt dissection through tissue, penetration into the thoracic cavity, dilation of a tract for tube placement, exploration of the thoracic cavity with a gloved finger, and finally insertion of a sterile tube into the intrathoracic space. The procedure is considered extremely painful despite the routine provision of systemic analgesics and local anesthetics.

Cadaver and animal studies have demonstrated the use of the Reactor chest tube device, a squeeze-activated thoracostomy trochar with placement of a clear sheath for chest tube insertion, to decrease procedure time, incision size, and blood loss. Case series and observational reports suggest lower rates of procedural complication and failure as well as increased patient satisfaction due to pain reduction.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects age ≥ 18 years old
2. Attending physician determination of need for urgent tube thoracostomy for treatment of traumatic pneumothorax, hemothorax, or hemopneumothorax.
3. Hemodynamically stable

Exclusion Criteria:

1. Pregnant patients
2. Prisoners
3. Need for emergency thoracostomy
4. Hemodynamic instability
5. Respiratory distress

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2019-07-01 (Estimated); Study Completion 2019-11-01 (Estimated)

PRIMARY OUTCOMES:
Patient report of pain | During procedure
  As measured on a 100mm VAS

SECONDARY OUTCOMES:
Procedure time | During procedure

IPD SHARING:
Plan to Share IPD: No